CLINICAL TRIAL: NCT04557995
Title: Efficacy and Safety of Erythrocytapheresis in Chronic Mountain Sickness: the ESCAPE-CMS Trial
Brief Title: Erythrocytapheresis for Chronic Mountain Sickness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ye Fan, Principal Investigator, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAP_2020
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Mountain Sickness
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erythrocytapheresis (Experimental): Erythrocytapheresis was was added to routine treatment
  Interventions: Procedure: Erythropheresis
- Routine treatment (No Intervention): Oxygen delivery and basic care

INTERVENTIONS:
Procedure: Erythropheresis — Draw blood from patient's vein and remove red blood cells as other components would be transfused back.
  Arms: Erythrocytapheresis

SUMMARY:
The clinical study is aimed to explore the efficacy and safety of erythrocytapheresis in chronic mountain sickness

DETAILED DESCRIPTION:
The clinical study is aimed to explore the efficacy and safety of erythrocytapheresis in chronic mountain sickness. People reside in highland diagnosed as chronic mountain sickness were included and randomly divided into two groups. In one group, routine therapy including oxygen inspiration would be performed, while in another erythropheresis would be added. Incremental shuttle walk test, symptom relief, and CMS score et al would be assessed and compared in the above two groups.

ELIGIBILITY:
Inclusion:

1. High-altitude residents or long-term dwellers (defined as continuous residence at ≥2,500 meters above sea level for ≥1 year), with no history of travel to low-altitude areas in the preceding 2 months and no planned travel to low-altitude areas during the study period;
2. Aged more than 18 years, any gender;
3. Diagnosed with CMS per the Qinghai CMS Criteria: Hemoglobin (Hb): Men: ≥210 g/L Women: ≥190 g/L At least one symptom/sign: headache, dizziness, dyspnea and/or palpitations, sleep disturbances, fatigue, localized cyanosis, burning sensation in palms/soles, venous dilatation, muscle/joint pain, loss of appetite, poor concentration or memory changes. CMS score ≥6;
4. Women of childbearing potential: negative pregnancy test (serum/urine) at screening. No pregnancy plans during the study period;
5. Willing to sign informed consent and able to comply with study procedures.

Exclusion:

1. Hematocrit <60%;
2. Patients with polycythemia due to: polycythemia vera, underlying cardiopulmonary diseases (e.g. COPD, chronic bronchitis, bronchiectasis, pulmonary fibrosis, heart disease), or other causes including malignancy;
3. Patients with active pneumonia, acute/chronic pulmonary embolism, or severe organ dysfunction (including cardiac, hepatic, or renal failure);
4. patients with contraindications to study procedures: erythrocytapheresis, pulmonary function tests, incremental shuttle walk test et al, including conditions such as pneumothorax, impaired consciousness, severe arrhythmia, or significant coagulation disorders et al.;
5. recent CMS-specific treatments (within the past 6 months): drug therapy, phlebotomy, or erythrocytapheresis;
6. pregnant or breastfeeding women;
7. current participation in other clinical trial (observational studies permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Incremental shuttle walk test | Within 48 hours after treatment is completed
  Measures the maximum distance a patient can walk at progressively increasing speeds until exhaustion, primarily assessing peak exercise capacity.
Chronic mountain sickness score | Within 48 hours after treatment is completed and during follow-up period
  A clinical tool used to assess the severity of chronic mountain sickness, also known as Monge's disease. It is based on symptoms and physiological markers related to excessive erythrocytosis (abnormally high red blood cell count) due to prolonged exposure to high altitude.

SECONDARY OUTCOMES:
SF-6D v2 score | Within 48 hours after treatment is completed and during follow-up period
  A preference-based health utility measure derived from the SF-36 or SF-12 health surveys. It is widely used in health economics and clinical research to assess health-related quality of life (HRQoL) and calculate Quality-Adjusted Life Years (QALYs) for cost-effectiveness analyses.
Blood oxygen saturation | Within 48 hours after treatment is completed and during follow-up period
  A measure of the percentage of hemoglobin binding sites in the bloodstream occupied by oxygen. It is a key indicator of respiratory and circulatory function, commonly assessed using a pulse oximeter (a non-invasive device that clips onto a finger, earlobe, or toe).

CONTACTS AND LOCATIONS:
Overall Officials: Ye Fan, Principal Investigator — Third Military Medical University
Locations (1):
- NO.953 Hospital, Xigazê, Tibet, China